CLINICAL TRIAL: NCT02590302
Title: Improving Transitions in Care for Children and Youth With Mental Health Concerns: Implementation and Evaluation of an Emergency Department Mental Health Clinical Pathway
Brief Title: Improving Transitions in Care for Children and Youth With Mental Health Concerns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Ministry of Health and Long Term Care (Other Government); Winchester District Memorial Hospital (Other); Queensway Carleton Hospital (Other); Youth Services Bureau (Unknown); Cornwall Community Hospital (Other)
Responsible Party: Principal Investigator, Mona Jabbour, Vice-Chief/Chair, Department of Pediatrics, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ChildrensHEO
Record Dates: First submitted 2015-10-20; First posted 2015-10-29 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Mental Health
Keywords: Clinical pathway; Mental Health; Emergency Department; Paediatric; Risk assessment; Service integration; Transitions in care; Implementation; Scoring tools; Clinical Pathway Evaluation
MeSH Terms: conditions — Psychological Well-Being; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dyads receiving the Implementation Phase (Other): Dyad 1 (CHEO-YSB) Dyad 2 (CGH-CCH) Dyad 3 (WDMH-CCH) Dyad 4 (QCH-YSB)
  Interventions: Other: Implementation Phase

INTERVENTIONS:
Other: Implementation Phase — Core Components of the implementation intervention include:
  * Hospital and CMHA project commitment
  * Site champion teams (from hospital and CMHA)
  * Memorandum of Agreement between Hospital and CMHA
  * Pre-intervention site visits
  * Education sessions
  * Posters/reminders
  * Instructional videos (HEADS ED video)
  Completed pathway implementation includes EDMHCP site-customization and committee approvals, consequent planning and agreements among ED-CMHA partners, delivery of at least two educational workshops, and EDMHCP availability in the ED. An 8-month period for EDMHCP implementation, with negotiated interim target dates was set for each site.

SUMMARY:
The overarching goal of this project is to improve timely access to appropriate mental health (MH) care for children and youth. The investigators will conduct and rigorously evaluate implementations of this pathway in four exemplar hospitals and associated CMHA dyads within a local health region. Outcomes-based validation of this pathway is important for effective adoption in other communities. A multiple baseline study design and conduct interrupted time-series analysis will be used to evaluate whether the EDMHCP has resulted in improved health care utilization, medical management, and health sector coordination. To ensure EDMHCP feasibility in various settings, implementation will occur in four exemplar hospital-community dyads with different workflows and patient populations.

DETAILED DESCRIPTION:
Commissioned by the Ontario Ministries of Health and Long Term Care(MOHLTC) and Child and Youth Services(MCYS), an expert-developed clinical pathway(CP) has been created with two main goals: 1) to guide risk assessment and disposition decision-making for children and youth presenting to the emergency department(ED) with MH concerns, and 2) to ensure seamless transition to follow-up services with community MH agencies(CMHAs) and providers. This pathway, referred to as the EDMHCP, is unique in undertaking to provide a seamless transition of care for children/youth and caregivers between hospital EDs and CMHAs.

Working with 4 exemplary hospital EDs and 2 Community Mental Health Agencies across Eastern Ontario, the investigators will conduct a 3-year mixed methods health services research project with three components to i) implement the EDMHCP using a theory driven, evidence-based approach, ii) evaluate EDMHCP effectiveness through measurement of relevant outcomes, and iii) conduct a process evaluation to document and assess the EDMHCP implementation strategy against the outcomes achieved.

This 3 year study will take place in five different phases, which include:

* Preparation: Qualitative interviews with ED team members and strategy development
* Implementation: Working with each ED team to implement the clinical pathway (including standardized assessments) within 8 months
* Post-implementation: Qualitative interviews with ED team members
* Data collection: 9-month pre/post chart audits of patients with mental health and caregiver satisfaction surveys
* Follow up: to discuss findings, database creation, and dissemination strategy.

To ensure the findings directly impact relevant service delivery areas, the investigators have specifically recruited study team members with decision-making authority and/or influence on delivery of care for children and youth with MH concerns. This project will provide an implementation model for the EDMHCP to be used in any ED and CMHA setting, and will demonstrate decreased wait times and increased access with EDMHCP adoption. The findings will guide policy decision-making on access to timely and appropriate MH care and add to current knowledge of implementation science. In addition to knowledge translation via team member dissemination within their areas of influence, the investigators plan to disseminate the findings through presentation at scientific and healthcare conferences, and publication in relevant peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 5.99 and < 18 years
* Presented to the ED of the four chosen hospitals within a selected 8 month time frame (between January, 2016 to May 2017)
* Mental health issue as their primary complaint (all complaints identified at triage as involving MH [psychosocial, emotional, behavioural])
* Proficient in English.

Exclusion Criteria:

* CTAS of 1 (Resuscitation)
* Patient is not medically stable
* Intubation/PICU care required
* Direct admission to hospital for ongoing medical management and observation
* Patients presenting with head injury or post-concussional syndrome

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3095 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving post-ED follow-up on the Services for Children and Adolescents Parent Interview questionnaire | 24 hours or 7 days
  The primary clinical outcome is the proportion of patients that receive the post ED follow-up as per the clinical pathway recommendations as measured by the Services for Children and Adolescents Parent Interview questionnaire
Proportion of patients with documented mental health recommendations in the medical chart | 24 hours or 7 days
  The primary process outcome is the proportion of patients with documented MH-specific recommendations (as defined by the project team) in the medical chart.

SECONDARY OUTCOMES:
Proportion of completed CP assessment forms filed in the health record to determine clinical pathway uptake in the Emergency Department | 9 months
  CP uptake in the ED will be measured through audits as the proportion of completed clinical pathway assessment forms filed in the health record
Patient perspectives of post-ED mental health service using The Services for Children and Adolescents-Parent Interview | 7-10 days
  Post ED uptake of recommended community MH services will be measured by The Services for Children and Adolescents-Parent Interview
Alignment of HEADS-ED assessment and mental health services | 7-10 days
  Alignment of recommended services documented in the patients health record (audit) to the HEADS-ED mental health screening tool assessment
Decreased length of stay | 26 months
  ED length of stay will be obtained from health record and NACRS administrative database
Patient satisfaction with ED visit measured by the Client Satisfaction Questionnaire | 7-10 days
  Patient/caregiver satisfaction with the ED visit will be measured by the Client Satisfaction Questionnaire
Decreased number of hospital admissions obtained from health record and NACRS administrative database | 26 months
  Hospital Admission will be obtained from health record and NACRS administrative database
Decreased number of ED Revisits from the health record and NACRS administrative database | 10 day and 3 months
  ED revisits will be obtained from the health record and NACRS administrative database

CONTACTS AND LOCATIONS:
Overall Officials: Mona Jabbour, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (2):
- Canada (2):
  - Children's Hopsital of Eastern Ontario, Ottawa, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario

REFERENCES:
- [Background] Cappelli M, Gray C, Zemek R, Cloutier P, Kennedy A, Glennie E, Doucet G, Lyons JS. The HEADS-ED: a rapid mental health screening tool for pediatric patients in the emergency department. Pediatrics. 2012 Aug;130(2):e321-7. doi: 10.1542/peds.2011-3798. Epub 2012 Jul 23. PMID 22826567
- [Background] Children's Hospital of Eastern Ontario. Advocacy Mental Health. Ottawa, Canada: http://www.cheo.on.ca/en/mentalhealth. Accessed August 22, 2014.
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Kataoka SH, Zhang L, Wells KB. Unmet need for mental health care among U.S. children: variation by ethnicity and insurance status. Am J Psychiatry. 2002 Sep;159(9):1548-55. doi: 10.1176/appi.ajp.159.9.1548. PMID 12202276
- [Background] Hacker K, Arsenault L, Franco I, Shaligram D, Sidor M, Olfson M, Goldstein J. Referral and follow-up after mental health screening in commercially insured adolescents. J Adolesc Health. 2014 Jul;55(1):17-23. doi: 10.1016/j.jadohealth.2013.12.012. Epub 2014 Feb 11. PMID 24525226
- [Background] Kirby, M.J.L., Keon, W.J. (2006). Out of the Shadows at Last: Transforming mental health, mental illness and addiction services in Canada. The Standing Senate Committee on Social Affairs, Science and Technology.
- [Background] Ontario Ministry of Health and Long-Term Care. Ontario's action plan for health care: Better patient care through better value from our health care dollars. Toronto, Canada: Government of Ontario; 2012. Available at: http://www.health.gov.on.ca/en/ms/ecfa/ healthy_change/docs/rep_healthychange.pdf. Accessed August 22, 2014.
- [Background] Ontario. Legislative Assembly. Select Committee on Mental Health and Addictions Final report, navigating the journey to wellness : the comprehensive mental health and addictions action plan for Ontarians; 2010 Available at: http://www.ontla.on.ca/committee-proceedings/committeereports/ files_pdf/Select%20Report%20ENG.pdf Accessed October 15, 2014.
- [Background] Provincial Council for Maternal and Child Health. Implementation Toolkit: Emergency Department Clinical Pathway for Children & Youth with Mental Health Conditions. Prov Counc Matern Child Heal. Available at: http://pcmch.on.ca/sites/default/files/Toolkit- ED_Clinical_Pathway-Tookit_ Sept_ 30_2013-FINAL_0.pdf. Accessed January 14, 2014.
- [Background] Open Minds, Healthy Minds. (2011). Ontario's comprehensive mental health and addictions strategy. Ottawa (ON): Government of Ontario. Available at: http://www.health.gov.on.ca/en/common/ministry/publications/reports/mental_health201 1/mentalhealth_rep2011.pdf Accessed October 15, 2014
- [Background] Bosch M, van der Weijden T, Wensing M, Grol R. Tailoring quality improvement interventions to identified barriers: a multiple case analysis. J Eval Clin Pract. 2007 Apr;13(2):161-8. doi: 10.1111/j.1365-2753.2006.00660.x. PMID 17378860
- [Background] Hartmann DP, Gottman JM, Jones RR, Gardner W, Kazdin AE, Vaught RS. Interrupted time-series analysis and its application to behavioral data. J Appl Behav Anal. 1980 Winter;13(4):543-59. doi: 10.1901/jaba.1980.13-543. PMID 16795632
- [Background] Jabbour M, Curran J, Scott SD, Guttman A, Rotter T, Ducharme FM, Lougheed MD, McNaughton-Filion ML, Newton A, Shafir M, Paprica A, Klassen T, Taljaard M, Grimshaw J, Johnson DW. Best strategies to implement clinical pathways in an emergency department setting: study protocol for a cluster randomized controlled trial. Implement Sci. 2013 May 22;8:55. doi: 10.1186/1748-5908-8-55. PMID 23692634
- [Background] Zhang F, Wagner AK, Soumerai SB, Ross-Degnan D. Methods for estimating confidence intervals in interrupted time series analyses of health interventions. J Clin Epidemiol. 2009 Feb;62(2):143-8. doi: 10.1016/j.jclinepi.2008.08.007. Epub 2008 Nov 17. PMID 19010644
- [Background] Wagner AK, Soumerai SB, Zhang F, Ross-Degnan D. Segmented regression analysis of interrupted time series studies in medication use research. J Clin Pharm Ther. 2002 Aug;27(4):299-309. doi: 10.1046/j.1365-2710.2002.00430.x. PMID 12174032
- [Background] Scott SD, Grimshaw J, Klassen TP, Nettel-Aguirre A, Johnson DW. Understanding implementation processes of clinical pathways and clinical practice guidelines in pediatric contexts: a study protocol. Implement Sci. 2011 Dec 28;6:133. doi: 10.1186/1748-5908-6-133. PMID 22204440
- [Background] Lougheed MD, Olajos-Clow J, Szpiro K, Moyse P, Julien B, Wang M, Day AG; Ontario Respiratory Outcomes Research Network. Multicentre evaluation of an emergency department asthma care pathway for adults. CJEM. 2009 May;11(3):215-29. doi: 10.1017/s1481803500011234. PMID 19523270
- [Background] Szpiro KA, Harrison MB, VanDenKerkhof EG, Lougheed MD. Asthma education delivered in an emergency department and an asthma education center: a feasibility study. Adv Emerg Nurs J. 2009 Jan-Mar;31(1):73-85. doi: 10.1097/TME.0b013e31818bf23d. PMID 20118856
- [Background] Bhogal S, Bourbeau J, McGillivray D, Benedetti A, Bartlett S, Ducharme F. Adherence to pediatric asthma guidelines in the emergency department: a survey of knowledge, attitudes and behaviour among health care professionals. Can Respir J. 2010 Jul-Aug;17(4):175-82. doi: 10.1155/2010/274865. PMID 20808976
- [Background] Michie S, Johnston M, Abraham C, Lawton R, Parker D, Walker A; "Psychological Theory" Group. Making psychological theory useful for implementing evidence based practice: a consensus approach. Qual Saf Health Care. 2005 Feb;14(1):26-33. doi: 10.1136/qshc.2004.011155. PMID 15692000
- [Background] Michie, S., Johnston, M., Harderman, W., & Eccles, M. (2008). From theory to intervention: Mapping theoretically derived behavioral determinants to behavior change techniques. Applied Psychology, 57(4), 660-680.
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Jensen PS, Eaton Hoagwood K, Roper M, Arnold LE, Odbert C, Crowe M, Molina BS, Hechtman L, Hinshaw SP, Hoza B, Newcorn J, Swanson J, Wells K. The services for children and adolescents-parent interview: development and performance characteristics. J Am Acad Child Adolesc Psychiatry. 2004 Nov;43(11):1334-44. doi: 10.1097/01.chi.0000139557.16830.4e. PMID 15502592
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] American Academy of Pediatrics; Committee on Pediatric Emergency Medicine; American College of Emergency Physicians; Pediatric Committee; Emergency Nurses Association Pediatric Committee. Joint policy statement--guidelines for care of children in the emergency department. Pediatrics. 2009 Oct;124(4):1233-43. doi: 10.1542/peds.2009-1807. Epub 2009 Sep 21. PMID 19770172
- [Background] Newton AS, Rathee S, Grewal S, Dow N, Rosychuk RJ. Children's Mental Health Visits to the Emergency Department: Factors Affecting Wait Times and Length of Stay. Emerg Med Int. 2014;2014:897904. doi: 10.1155/2014/897904. Epub 2014 Jan 19. PMID 24563785
- [Background] Newton, A. S., Rosychuk, R. J., Ali, S., Cawthorpe, D., Curran, J., Dong, K., … Urichuk, L. (2011). The Emergency Department Compass: Children's Mental Health. Pediatric mental health emergencies in Alberta, Canada: Emergency department visits by children and youth aged 0 to 17 years, 2002-2008. Edmonton, AB.
- [Background] Chandra A, Minkovitz CS. Stigma starts early: gender differences in teen willingness to use mental health services. J Adolesc Health. 2006 Jun;38(6):754.e1-8. doi: 10.1016/j.jadohealth.2005.08.011. PMID 16730608
- [Derived] Tucci A, Cloutier P, Polihronis C, Kennedy A, Zemek R, Gray C, Reid S, Pajer K, Gardner W, Barrowman N, Cappelli M, Jabbour M. Improving transitions in care for children and youth with mental health concerns: implementation and evaluation of an emergency department mental health clinical pathway. BMC Health Serv Res. 2025 Mar 31;25(1):475. doi: 10.1186/s12913-025-12524-z. PMID 40165260
- [Derived] Jabbour M, Reid S, Polihronis C, Cloutier P, Gardner W, Kennedy A, Gray C, Zemek R, Pajer K, Barrowman N, Cappelli M. Improving mental health care transitions for children and youth: a protocol to implement and evaluate an emergency department clinical pathway. Implement Sci. 2016 Jul 7;11(1):90. doi: 10.1186/s13012-016-0456-9. PMID 27389410